CLINICAL TRIAL: NCT06777511
Title: Advancing Antimicrobial Photodynamic Therapy to Prevent Infection in Osseointegrated Prosthesis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief, Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02003108
Record Dates: First submitted 2025-01-08; First posted 2025-01-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Amputation; Osseointegration
MeSH Terms: interventions — Aminolevulinic Acid; Photochemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — swab specimens of the stoma site, collected for determining bacterial bioburden
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Osseointegration patients: All patients >18 years with osseointegrated prostheses.
  Interventions: Drug: 5-aminolevulinic acid (5-ALA); Device: Photodynamic therapy (PDT)

INTERVENTIONS:
Drug: 5-aminolevulinic acid (5-ALA) — All patients who are recruited and enrolled into this study use topical 5- ALA, in combination with the light delivery device as part of their standard stoma management.
Device: Photodynamic therapy (PDT) — All patients who are recruited and enrolled into this study use topical 5- ALA, in combination with the light delivery device photodynamic therapy device as part of their standard stoma management.

SUMMARY:
This will be a prospective observational trial enrolling 20 patients with osseointegrated prostheses. Participants will be recruited from the orthopaedic outpatient clinic at Walter Reed National Military Medical Center in Bethesda, MD.

All eligible consenting patients will undergo daily stoma management per standard of care.

Patients will integrate antimicrobial photodynamic therapy into their stoma management program. The first treatment will take place in the orthopaedic clinic. All others will take place at home. Topical 5-ALA will be applied to the metal at the penetration site. After 2 hours, the light delivery device will be utilized and light will be administered for 15 minutes.

Data collection: After obtaining informed consent, study personnel will record injury-specific variables, surgery-specific variables, other variables related to their hospital course, demographic variables as well as comorbidities on the study case report forms (CRFs). They will obtain this information directly from the participant, from the participant's medical record, and the participant's treating orthopaedic surgeon or other health care providers. Baseline data collection points include participant characteristics and amputation details such as age, sex, comorbidities, highest education level achieved, social support, initial reason for amputation, type of amputation and all surgical dates. Study participants will be followed at 1 and 2 weeks after initiation of PDT treatment. To ensure research participant safety, serious adverse events (SAEs) will be documented and promptly submitted to the local IRB as per the required reporting processes.

Follow-up: Study participants will be followed at 1 week and 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients with osseointegrated prostheses 18 years of age or older

Exclusion Criteria:

* Ongoing infection
* Pregnant
* Anticipated issues with compliance or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years with osseointegrated prostheses are eligible. Patients will be excluded if they have an ongoing infection, are pregnant or if it is anticipate that they will have issues with compliance or follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 2 weeks
  Feasibility will be defined as 80% of patients successfully completing the administration protocol as well as 1 week/2-week follow-up.

SECONDARY OUTCOMES:
Treatment Evaluation Inventory-Short Form (TEI-SF) | 2 weeks
  The TEI-sf is a 9-item questionnaire used to measure intervention acceptability from the participants point of view. Scores range from 9 to 45, and scores above 27 are considered acceptable.
System Usability Scale (SUS) | 2 weeks
  The SUS is a reliable 10-item usability measure with scores that range from 0 to 100 (an above average score is 68 or higher.
Bioburden quantification (16S rRNA sequencing) | 2 weeks
  Bioburden will be quantified using quantitative PCR-based assays as well as addition of a "spikein" of a defined quantity of bacterial cells derived from halophilic organism Salnibacter ruber.
Bioburden quantification (Optical Coherence Tomography (OCT) | 2 weeks
  Biofilm will be imaged and quantified on the metal abutment
OCT "virtual biopsy" | 2 weeks
  Presence of inflammation, hypergranulation, and any resulting changes (e.g., the degree of epidermal regression, dermal attachment to the implant, and epithelial layer thickness) can be quantified through morphologic analysis of the OCT B-scans. Scars are characterized by excessive collagen deposition, increased blood vessel density, and parallel blood vessel organization compared with normal skin.
Scar thickness | 2 weeks
  Scar thickness measured using OCT
Blood vessel density | 2 weeks
  Blood vessel density measuring using OCT
Presence of hypergranulation | 2 weeks
  Hypergranulation measured using OCT
Pain during light exposure | 2 weeks
  Patient reported pain during light exposure
Discomfort, burning, itchiness, or redness | 2 weeks
  Patient reported discomfort, burning, itchiness or redness

IPD SHARING:
Plan to Share IPD: No